CLINICAL TRIAL: NCT03894462
Title: Effectiveness of a Targeted Brief Intervention for Recent Suicide Attempt Survivors
Brief Title: Study About Treatment After a Suicide Attempt
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Northwestern University (Other); Hutchings Psychiatric Center (Unknown); University of Arkansas (Other); State University of New York - Upstate Medical University (Other)
Responsible Party: Principal Investigator, Anthony Pisani, Principal Investigator, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 3353
Record Dates: First submitted 2019-02-12; First posted 2019-03-28 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2024-10

CONDITIONS: Suicide, Attempted
Keywords: Zero Suicide; Effectiveness; Brief Treatment; Interpersonal Theory; Cost-Effectiveness
MeSH Terms: conditions — Suicide, Attempted

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Care Provider
Masking Description: We do not inform providers giving usual care whether their patients are receiving ASSIP. However, providers may find out through ordinary course of usual care being provided.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Zero Suicide Usual Care (Active Comparator): In Onondaga County, New York State (NYS) aims to implement a countywide "Zero Suicide Safety Net" of providers who share enhanced protocols for clinical care, staff training, and data collection (improved coding of suicidal behavior). Participating behavioral health systems have agreed to common protocols for clinical care, training, and data collection. Participating providers receive robust training in suicide prevention best practices. Because of the wide participation of mental health facilities in the NYS Office of Mental Health (OMH) Zero Suicide project, most subjects who engage in outpatient treatment will receive that treatment in facilities that are adopting NYS Zero Suicide protocols. Those who do not engage in care will nonetheless experience enhanced transition and follow-up contact from the services from which they are discharged.
  Interventions: Behavioral: Zero Suicide Usual Care
- Zero Suicide Usual Care + ASSIP (Experimental): Patients in this treatment arm will receive ASSIP brief therapy in addition to being able to access any usual care as recommended by their provider.
  ASSIP is a manualized, three-session intervention, delivered either in-person or via telehealth: In Session 1, the therapist guides the patient in telling the story of their attempt. The session is video recorded. In Session 2, the therapist and patient sit side-by-side to view selections of the video, working together to understand the feelings and events that preceded the attempt. The patient is assigned a homework task. In Session 3, the therapist and patient create a summary of the suicide attempt and what led up to it, along with creating a personal safety plan.
  Interventions: Behavioral: Attempted Suicide Short Intervention Program

INTERVENTIONS:
Behavioral: Attempted Suicide Short Intervention Program — ASSIP is a manualized, three-session intervention, delivered either in-person or via telehealth: In Session 1, the therapist guides the patient in telling the story of their attempt. The session is video recorded. In Session 2, the therapist and patient sit side-by-side to view selections of the video, working together to understand the feelings and events that preceded the attempt. The patient is assigned a homework task. In Session 3, the therapist and patient create a summary of the suicide attempt and what led up to it, along with creating a personal safety plan.
  Arms: Zero Suicide Usual Care + ASSIP
Behavioral: Zero Suicide Usual Care — Participants will have access to outpatient treatment in facilities that are adopting NYS Zero Suicide protocols. Those who do not engage in care will nonetheless experience enhanced transition and follow-up contact from the services from which they are discharged.
  Arms: Zero Suicide Usual Care

SUMMARY:
Effective, brief, low-cost interventions for individuals who attempt suicide are needed to save lives and achieve the goals of the National Strategy for Suicide Prevention. In response to a National Institute for Mental Health (NIMH) Notice of Interest, this time-sensitive proposal leverages an existing federal investment in Zero Suicide to test the effectiveness of a highly promising new treatment for recent suicide attempt survivors and learn how it works. If hypotheses are supported, the study will provide evidence of a brief, practical, and cost-effective therapy that reduces suicide reattempts in a real-world health setting.

DETAILED DESCRIPTION:
Suicide rates are rising in the US and more than a million Americans try to take their own lives each year. Effective, brief, low-cost interventions for individuals who attempt suicide are essential to saving lives and achieving the goals of the National Strategy for Suicide Prevention. This study takes advantage of a time-sensitive research opportunity to test the effectiveness of the Attempted Suicide Short Intervention Program (ASSIP), a manualized 3-session intervention for recent suicide attempt survivors that produced dramatic reductions in suicide attempts in a efficacy trial-80% fewer reattempts and an average of 72% fewer hospital days over 24 months in the intervention group compared to controls. This research will now test its effectiveness of in the US public mental health care system, examine theoretically grounded mechanisms, and explore cost-effectiveness. ASSIP is currently being implemented by New York State in a Zero Suicide initiative funded by SAMHSA. Consistent with NIMH Notice of Interest MH-17-03, this project leverages this federal investment and a strong state partnership to conduct effectiveness research.

Effectiveness. The primary aim of this study is to determine the effectiveness of ASSIP in reducing suicide reattempts in a community mental health setting in the U.S. To accomplish this aim the investigators will conduct a randomized controlled trial with 400 individuals referred from psychiatric inpatient and emergency services following a suicide attempt. Participants will be randomized to receive either usual care + ASSIP (intervention arm) or usual care only (control arm), and followed for assessments at baseline, 6-weeks 3-, 6-, 12-, and 18-months.

Mechanism. The secondary aim of this study to examine the psychological mechanisms of ASSIP, as predicted by the Interpersonal Theory of Suicide. To accomplish this aim the investigators will conduct statistical analyses of a mediation model to determine (a) whether ASSIP improves perceptions of low belonging and being a burden on others, and (b) whether the effect of treatment on reductions in suicide re-attempts is mediated by these improvements.

Cost-Effectiveness. The exploratory aim is to identify potential implementation costs, barriers, and facilitators for delivering ASSIP. A stakeholder summary report will be written and disseminated, including an estimate, from the perspective of an ASSIP provider, the incremental cost per suicide attempt averted by delivering ASSIP to supplement usual care following a suicide attempt. This report can be used by organizations and localities considering implementing ASSIP as part of their Zero Suicide strategy.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years or older.
2. Suicide attempt within the past 60 days defined by intent to die using a standard item.
3. Ability and willingness to provide information and permission to contact at least one person in the case of a need to contact them to promote subject safety or inability to reach the subject for follow-up.

Exclusion Criteria:

1. Acute psychiatric instability (e.g., psychotic symptoms).
2. Inability to communicate in English (ASSIP is only provided by the clinic in English).
3. Residing outside of NYS (during the period eligible for ASSIP)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 443 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Time to Suicide Attempt | Up to 18 months
  Time from randomization to first suicide re-attempt

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Rochester Medical Center, Rochester, New York
  - St. Joseph's Health Hospital, Syracuse, New York
  - Upstate University Hospital, Syracuse, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gysin-Maillart A, Schwab S, Soravia L, Megert M, Michel K. A Novel Brief Therapy for Patients Who Attempt Suicide: A 24-months Follow-Up Randomized Controlled Study of the Attempted Suicide Short Intervention Program (ASSIP). PLoS Med. 2016 Mar 1;13(3):e1001968. doi: 10.1371/journal.pmed.1001968. eCollection 2016 Mar. PMID 26930055
- [Derived] Pisani A, Connor K, Van Orden K, Jordan N, Landes S, Curran G, McDermott M, Ertefaie A, Kelberman C, Ramanathan S, Carruthers J, Mossgraber K, Goldston D. Effectiveness of a targeted brief intervention for recent suicide attempt survivors: a randomised controlled trial protocol. BMJ Open. 2023 Mar 3;13(3):e070105. doi: 10.1136/bmjopen-2022-070105. PMID 36868590
- [Derived] Witt KG, Hetrick SE, Rajaram G, Hazell P, Taylor Salisbury TL, Townsend E, Hawton K. Psychosocial interventions for self-harm in adults. Cochrane Database Syst Rev. 2021 Apr 22;4(4):CD013668. doi: 10.1002/14651858.CD013668.pub2. PMID 33884617